CLINICAL TRIAL: NCT02240888
Title: Vaccination in Inflammatory Rheumatic Disease (VACCIMIL). The Impact of Antirheumatic Treatment on Antibody Response
Acronym: Vaccimil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, meliha crnkic kapetanovic, MD, PhD, associate professor, Region Skane
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/341; Vaccimil (Other: Vaccimil)
Record Dates: First submitted 2014-09-04; First posted 2014-09-16 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: RA; SLE; Vasculitis; Scleroderma; Sjögrens; Syndrome
Keywords: pneumococcal; vaccination; antibody; response; immunosuppressive; treatment; inflammatory; rheumatic; disease
MeSH Terms: conditions — Vasculitis; Scleroderma, Diffuse; Syndrome; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- vaccinated patients (Active Comparator): patients with different inflammatory rheumatic disease immunized with 0,5 mg pneumococcal conjugate vaccine i.m.
  Interventions: Biological: 0,5 mg Prevenar i.m.; Biological: 0,5 mg seasonal influenza vaccine i.m.
- vaccinated controls (Active Comparator): healthy controls immunized with 0,5 mg pneumococcal conjugate vaccine i.m.
  Interventions: Biological: 0,5 mg Prevenar i.m.; Biological: 0,5 mg seasonal influenza vaccine i.m.
- seasonal influenza vaccine (Active Comparator): patients with different inflammatory rheumatic diseases immunized with 0,5 mg seasonal influenza vaccine i.m.
  Interventions: Biological: 0,5 mg Prevenar i.m.; Biological: 0,5 mg seasonal influenza vaccine i.m.
- non-vaccinated controls (Active Comparator): healthy controls immunized with 0,5 mg seasonal influenza vaccine i.m.
  Interventions: Biological: 0,5 mg Prevenar i.m.; Biological: 0,5 mg seasonal influenza vaccine i.m.

INTERVENTIONS:
Biological: 0,5 mg Prevenar i.m.
Biological: 0,5 mg seasonal influenza vaccine i.m.

SUMMARY:
The overall objective of this project is to study the influence of modern anti-inflammatory treatments in established inflammatory rheumatic diseases (IRD) on immune response elicited by pneumococcal vaccination using 13-valent conjugate vaccine and influenza vaccination. In addition, the aim is to study the clinical aspects of vaccination regarding: tolerability in immunosuppressed patients with IRD, impact on existing rheumatic disease, possible association with onset of new autoimmune diseases, long-term immunity following pneumococcal vaccination, efficacy in preventing invasive pneumococcal diseases and influenza related serious infections. Results from this study are expected to bridge the existing knowledge gap and contribute to body of evidence needed for recommendations and implementation of vaccination program in IRD patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with IRD receiving active anti-rheumatic treatments with DMARDs or biological remedies are offered to participate in the study. The protocol permits stratification for prednisolone usage, smoking habits and alcohol consumption.

Exclusion Criteria:

* age <18 years;
* pregnancy,
* known intolerance of vaccine,
* ongoing infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-10; Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
antibody response following vaccination | 4-6 weeks after pneumococcal and influenza vaccination
  measurement of antibody levels against different pneumococcal capsular serotypes and 3 influenza virus strains

SECONDARY OUTCOMES:
long-term immunity following pneumococcal vaccination | 3 years after pneumococcal vaccination
  measurement of antibody levels against different pneumococcal capsular serotypes
long-term immunity after vaccination with pneumococcal conjugate vaccine | 5 years after vaccination
  measurement of antibody levels against different pneumococcal polysaccharide serotypes

OTHER OUTCOMES:
The occurence of severe pneumococcal infections in immunized patients | within 5 years after pneumococcal vaccination
  Analysis of the occurence of severe pneumococcal infections in immunized patients compared to matched not-immunized controls

CONTACTS AND LOCATIONS:
Overall Officials: Meliha C Kapetanovic, MD, PhD, Principal Investigator — Region Skåne; Jehns Martineus, MD, Study Director — Skåne Universitets sjukhus, dept of rheumatology
Locations (1):
- Skåne University hospital, Dept of rheumatology, Lund, Sweden

REFERENCES:
- [Derived] Nived P, Saxne T, Geborek P, Mandl T, Skattum L, Kapetanovic MC. Antibody response to 13-valent pneumococcal conjugate vaccine is not impaired in patients with rheumatoid arthritis or primary Sjogren's syndrome without disease modifying treatment. BMC Rheumatol. 2018 Apr 5;2:12. doi: 10.1186/s41927-018-0019-6. eCollection 2018. PMID 30886963
- [Derived] Hesselstrand R, Nagel J, Saxne T, Geborek P, Skattum L, Kapetanovic MC. Immunogenicity and safety of pneumococcal vaccination in patients with systemic sclerosis. Rheumatology (Oxford). 2018 Apr 1;57(4):625-630. doi: 10.1093/rheumatology/kex471. PMID 29325173
- [Derived] Nived P, Nagel J, Saxne T, Geborek P, Jonsson G, Skattum L, Kapetanovic MC. Immune response to pneumococcal conjugate vaccine in patients with systemic vasculitis receiving standard of care therapy. Vaccine. 2017 Jun 22;35(29):3639-3646. doi: 10.1016/j.vaccine.2017.05.044. Epub 2017 May 25. PMID 28552512
- [Derived] Kapetanovic MC, Nagel J, Nordstrom I, Saxne T, Geborek P, Rudin A. Methotrexate reduces vaccine-specific immunoglobulin levels but not numbers of circulating antibody-producing B cells in rheumatoid arthritis after vaccination with a conjugate pneumococcal vaccine. Vaccine. 2017 Feb 7;35(6):903-908. doi: 10.1016/j.vaccine.2016.12.068. Epub 2017 Jan 9. PMID 28081972